CLINICAL TRIAL: NCT06593470
Title: Mindfulness-Based Substance Use Prevention (MINDS-UP): a Randomized Controlled Trial
Brief Title: Mindfulness-Based Substance Use Prevention (MINDS-UP)
Acronym: MINDS-UP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, David Saunders, MD PhD, Assistant Prof of Psychiatry, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: #Pro00076319; K12DA000357 (NIH)
Record Dates: First submitted 2024-08-15; First posted 2024-09-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Substance Use
MeSH Terms: conditions — Substance-Related Disorders | interventions — Health; Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Sport: Prevention Plus Wellness (PPW) (Active Comparator): Sport: Prevention Plus Wellness (PPW) is a brief, evidence-based substance use prevention program for youth. PPW consists of a single remote-delivered 45-minute session by a research assistant (RA) trained in PPW that is interactive and intended for use by youth in the home setting. It involves screening youth to increase awareness of their current health behaviors; motivational enhancement for change; and establishing a behavior goal plan.
  Interventions: Behavioral: Prevention Plus Wellness
- MINDS-UP with MRI + PPW (Experimental): MINDS-UP consists of 4 x 60-minute sessions, once weekly over 4 weeks. MINDS-UP will be delivered to participants remotely, in a 1:1 setting, taught by the meditation teachers that will be hired and trained by Dr. Saunders. Additionally, participants will be provided audio files of 5-10-minute guided meditation practices, led by Dr. Saunders, as homework. Half of those randomized to receive MINDS-UP + PPW (n=10) will receive functional and structural MRI before and after MINDS-UP to evaluate feasibility and acceptability of our MRI procedures and study design. Participants randomized to MINDS-UP with MRI arm will also complete PPW.
  Interventions: Behavioral: MINDS-UP; Behavioral: Prevention Plus Wellness; Diagnostic Test: fMRI
- MINDS-UP without MRI + PPW (Experimental): MINDS-UP consists of 4 x 60-minute sessions, once weekly over 4 weeks. MINDS-UP will be delivered to participants remotely, in a 1:1 setting, taught by the meditation teachers that will be hired and trained by Dr. Saunders. Additionally, participants will be provided audio files of 5-10-minute guided meditation practices, led by Dr. Saunders, as homework. Participants randomized to MINDS-UP without MRI arm will also complete PPW.
  Interventions: Behavioral: MINDS-UP; Behavioral: Prevention Plus Wellness

INTERVENTIONS:
Behavioral: MINDS-UP — MINDS-UP is a substance use prevention program for children/adolescents.It consists of 4 x 60-minute sessions, once weekly over 4 weeks. The four MINDS-UP classes will focus on the following: Mindfulness of Body; Mindfulness of Mind; Mindfulness of Environment/Community; Kindness, Compassion, Joy and Equanimity, respectively.
  Arms: MINDS-UP with MRI + PPW; MINDS-UP without MRI + PPW
Behavioral: Prevention Plus Wellness — PPW is a standardized, empirically-based intervention for substance use prevention in adolescents ages 10-14. It consists of 1 45-60 minute session between an adolescent and a trained PPW teacher.
  Other Names: PPW
Diagnostic Test: fMRI — Functional MRI to investigate preliminary neural mechanisms of MINDS-UP
  Arms: MINDS-UP with MRI + PPW

SUMMARY:
The goal of this clinical trial is to test the feasibility, behavioral/neural mechanisms, and preliminary efficacy of "MINDfulness-based Substance Use Prevention Program," or "MINDS-UP", a novel substance use prevention meditation intervention for children and adolescents between the ages of 10 and 14. The main questions it aims to answer are:

1. Is MINDS-UP feasible and what is its preliminary efficacy?
2. Are MRI protocol and procedures feasible?

An additional exploratory question is:

Are there neural and psychopathological mechanisms through which MINDS-UP might work?

Researchers will compare Sport - Prevention Plus Wellness (PPW) (an evidence based substance use prevention program) to Sport - Prevention Plus Wellness + MINDS-UP to examine the preliminary efficacy of MINDS-UP.

Participants will

* take assessment #1
* have 2 MRIs and take MINDS-UP, just take MINDS-UP or have a delayed start
* take assessment #2
* take PPW, a single remote and research assistant-delivered 45-minute session
* take assessment #3
* take assessment #4

ELIGIBILITY:
Inclusion Criteria:

* Youth is ages 10-14 years on the day of screening [i.e., does not turn 15 before or on the day of screening]
* Access to a smart phone, tablet, or computer with Wi-Fi
* English-speaking

Exclusion Criteria:

* Has been diagnosed with or received treatment for one of the following mental health problems: depression, bipolar disorder, schizophrenia, autism spectrum disorder, intellectual disability, or substance use disorder.
* Youth is actively involved in another Boricua Youth Study (BYS)
* Youth's sibling is or has previously been enrolled in MINDS-UP.

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 45 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Teacher Rated Participation | Completion of Study (up to 36 months)
  Research Assessment Package for Schools - Teacher Rated
Acceptability | Completion of Study (up to 36 months)
  Acceptability of Intervention Measure
Retention | Completion of Study (up to 36 months)
  Percent of participants who completed all study procedures among those who were randomized
Attendance | Completion of Study (up to 36 months)
  Percent of scheduled sessions that were completed by the participant.
Homework Completion | Completion of Study (up to 36 months)
  Percentage of assigned homeworks that were completed by the participant.
Participation (student) | Completion of Study (up to 36 months)
  Research Assessment Package for Schools - Student Engagement

SECONDARY OUTCOMES:
MRI retention | Completion of Study (up to 36 months)
  Percentage of participants randomized to receive MRI that complete both MRIs
Future MRI endorsement | Completion of Study (up to 36 months)
  Percentage of participants who endorse willingness to undergo a future research MRI scan
Anxiety and Depression | 4-6 weeks, 6 months, and 12 months
  Pre-assessment to post-assessment (and 6 and 12 month-follow-up) difference in score on the Revised Childhood Anxiety and Depression scale, a 47-item self-report scale that assesses childhood/adolescent anxiety and depression symptoms across six sub-domains.
Mindfulness | 4-6 weeks, 6 months, and 12 months
  Pre-assessment to post-assessment (and 6- and 12-month follow-up) difference in score on the Child and Adolescent Mindfulness Measure (CAMM); the CAMM is a 10-item measure of self-reported mindfulness; scores range from 0 to 40, with higher scores indicating higher mindfulness
Externalizing Problems (parent-report) | 4-6 weeks, 6 months, and 12 months
  Pre-assessment to post-assessment (and 6- and 12-month follow-up) difference in score on the externalizing problems subscale on the Child Behavior Checklist (CBCL), which is comprised of 33 questions; individual item scores range from 0 to 2; higher scores indicate higher amount of externalizing problems
Externalizing Problems (self-report) | 4-6 weeks, 6 months, and 12 months
  Pre-assessment to post-assessment (and 6- and 12-month follow-up) difference in the total score on the externalizing problems subscale on the Youth Self Report, which is comprised of 112 questions; individual item scores range from 0 to 2; higher scores indicate higher amount of behavioral problems
Total Problems (self-report) | 4-6 weeks, 6 months, and 12 months
  Pre-assessment to post-assessment (and 6- and 12-month follow-up) difference in the total score on the total problems subscale Youth Self Report; the survey is comprised of 112 items, with individual item scores range from 0 to 2; higher scores indicate higher amount of behavioral problems
Total Problems (parent-report) | 4-6 weeks, 6 months, and 12 months
  Pre-assessment to post-assessment (and 6- and 12-month follow-up) difference in the total score on the total problems subscale on the Child Behavior Checklist (CBCL), which is comprised of 98 questions; individual item scores range from 0 to 2; higher scores indicate higher amount of behavioral problems
Cannabis Use | 4-6 weeks, 6 months, and 12 months
  Cannabis use as measured by the Marijuana Low-Level Use Measure, a short tool that measures early/first use of cannabis.
Alcohol sipping | 4-6 weeks, 6 months, and 12 months
  Low-level and early alcohol use as characterized by the iSay Sipping Inventory. This survey characterizes low level and first/early alcohol use, including age at first sip, whether that drink was completed, and behaviors after the first sip.
Tobacco Use | 4-6 weeks, 6 months, and 12 months
  Tobacco use as measured by Tobacco Low Level Use Measure. This is a short tool that measures number of times used, type of tobacco/nicotine used, duration of use, and frequency of use.
ADHD Symptoms | 4-6 weeks, 6 months, and 12 months
  Pre-assessment to post-assessment (and 6- and 12-month follow-up) difference in score on the externalizing problems subscale on the Child Behavior Checklist (CBCL), which is comprised of 33 questions; individual item scores range from 0 to 2; higher scores indicate higher amount of externalizing problems

IPD SHARING:
Plan to Share IPD: No